CLINICAL TRIAL: NCT01710904
Title: The Evaluation of Targinact® in Daily Practice, With Regards to Pain Relief and Constipation, in Chronic Severe Pain Patients Compared to Previous Prolonged Release Oxycodone Treatment: a Non-interventional, Observational Study.
Brief Title: A Non-interventional, Observational Study for Targinact® Treatment in Patients With Chronic Severe Pain
Status: Completed | Type: Observational
Sponsor: Mundipharma CVA (Other)
Responsible Party: Sponsor
Other Study IDs: OXN9511
Record Dates: First submitted 2012-10-16; First posted 2012-10-19 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Severe Pain
Keywords: Chronic pain; Severe pain; Oxycodone; Naloxone; Opioid-induced constipation; Opioid; Quality of life; Laxative; Analgesic rescue medication
MeSH Terms: conditions — Chronic Pain; Pain; Opioid-Induced Constipation | interventions — oxycodone naloxone combination; Oxycodone; Naloxone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Targinact® (oxycodone/naloxone)

SUMMARY:
This non-interventional, observational study is set up on request of the Belgian reimbursement authorities and evaluates the efficacy of Targinact with regard to pain relief and constipation in daily clinical practice in Belgium compared to the previous analgesic treatment with prolonged release oxycodone. Only patients eligible for Targinact® reimbursement in Belgium are included.

DETAILED DESCRIPTION:
Patients are treated with Targinact® according to daily clinical practice during at least 12 weeks and are monitored during study 3 visits. Parameters assessed are pain relief, constipation, use of laxatives, use of analgesic rescue medication, use of concomitant medication, quality of life and safety of Targinact® treatment. These parameters, except for safety assessment, are compared between Targinact® treatment and previous analgesic treatment with prolonged release oxycodone.

ELIGIBILITY:
Inclusion criteria: patients included are patients who

* are eligible for Targinact® treatment according to the Targinact® SPC AND
* who have previously been treated with PR oxycodone during at least the last 30 days before study inclusion AND
* who are constipated (BFI > 30) AND
* have used at least 2 laxatives with different modes of action during the previous PR oxycodone treatment

Exclusion criteria are based on Targinact® SPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary and Secondary Care
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of responders after Targinact treatment compared to the previous treatment with prolonged release oxycodone. | 12 weeks
  A responder is defined as a patient who shows no worsening of pain (pain score has increased ≤ 1 unit on a 11-points pain NRS) at V3/the last visit compared to V1 or has a NRS ≤4 on a 11-points pain NRS at V3/the last visit AND has a reduction in BFI ≥ 12 units at V3/the last visit compared to V1 or has a BFI ≤30 at V3/ the last visit.

SECONDARY OUTCOMES:
To assess laxative use during Targinact® treatment compared to previous PR oxycodone treatment (by physician) | 12 weeks
  To assess laxative use during Targinact® treatment compared to previous PR oxycodone treatment (by physician)
To assess the use of analgesic rescue medication during Targinact® treatment compared to previous PR oxycodone treatment (by physician) | 12 weeks
  To assess the use of analgesic rescue medication during Targinact® treatment compared to previous PR oxycodone treatment (by physician)
To evaluate the quality of life (EQ-5D questionnaire) during Targinact® treatment compared to previous PR oxycodone treatment (by patient) | 12 weeks
  To evaluate the quality of life (EQ-5D questionnaire) during Targinact® treatment compared to previous PR oxycodone treatment (by patient)
To assess safety of Targinact® treatment (by physician) | 12 weeks
  Safety will be assessed by documentation of adverse events, collected via spontaneous reports and patient documentation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Brussels, Brussels, Belgium

REFERENCES:
- See also: Clinical Therapeutics — http://dx.doi.org/10.1016/j.clinthera.2015.02.010